CLINICAL TRIAL: NCT00252148
Title: Randomized, Placebo-Controlled, Dose-Escalating, Double-Blinded Phase 1 Safety and Immunogenicity Study of a Modified Vaccinia Ankara (MVA) Vectored HIV-1 (ADMVA) Vaccine Administered Intramuscularly to HIV-Uninfected, Healthy Volunteers
Brief Title: Safety and Immunogenicity of a Modified Vaccinia Ankara (MVA) HIV Vaccine in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Aaron Diamond AIDS Research Center (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI C002
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infection
Keywords: HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADMVA (Active Comparator): ADMVA dosage escalation
  Interventions: Biological: ADMVA
- Placebo (Placebo Comparator): Placebo is 10mM TRIS HCl, 140mM NaCl, ph 7.7
  Interventions: Biological: ADMVA

INTERVENTIONS:
Biological: ADMVA — experimental HIV vaccine, MVA vector expressing HIV clade C env, gag, pol, nef, and tat

SUMMARY:
The purpose of this study is to determine the safety of an immune response to an investigational HIV vaccine, ADMVA, at three different dosage levels, in adults who are not infected with HIV

DETAILED DESCRIPTION:
This is a dose escalation trial. Study site staff and volunteers will be blinded. Blinding will not apply to the assignment of dose levels (low, middle or high).

Volunteers will be screened up to 42 days before enrolment and will be followed for 18 months after the first vaccination.

16 volunteers will be randomized in a 3:1 ratio of active vaccine to placebo. Safety and tolerability of the ADMVA vaccine/placebo will be evaluated at least 14 days after the 12th volunteer in the low dose group receives the second injection before proceeding to the middle dose group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females, as assessed by a medical history, physical exam, and laboratory tests;
* Age of at least 18 years of age on the day of screening and no greater than 40 years on the day of first vaccination;
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 18 months);
* In the opinion of the principal investigator or designee has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed;
* Willing to undergo HIV Testing and counseling, and receive HIV test results;
* If sexually active female, using an effective method of contraception from screening until at least 4 months after last vaccination. All female volunteers must be willing to undergo urine pregnancy tests.
* If sexually active male, willing to use an effective method of contraception from screening until 4 months after the last vaccination and will be advised not to get his partner pregnant.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection;
* Reported high-risk behavior for HIV infection defined as:

Within 6 months before vaccination, the volunteer has:

* Had unprotected vaginal or anal sex with a known HIV infected person or with a casual partner.
* Engaged in sex work for money or drugs
* Used injection drugs (illicit), or
* Acquired an STD;
* Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, antiviral, anticancer, or other medications considered significant by the trial physician within the last 6 months;
* Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation;
* Any of the following abnormal laboratory parameters listed below:
* Hemoglobin: <9.0 g/dL
* Absolute Neutrophil Count (ANL): ≤ 999/mm3
* Absolute Lymphocyte Count (ALC): ≤ 500/mm3
* Platelets: ≤ 90,000 ≥ 550,000/mm3
* Creatinine: > 1.4 x ULN
* AST: >3.0 x ULN
* ALT: >3.0 x ULN
* Urine dipstick: blood = 2+ or more (except in menstruating females); protein = 2+or more
* Cardiac troponin I: > ULN;
* Confirmed diagnosis of hepatitis B (surface antigen, HbsAg); hepatitis C (HCV antibodies) or active syphilis;
* If female, pregnant or planning a pregnancy within 4 months after last vaccination or lactating;
* Receipt of a live attenuated vaccine (other than influenza) within 30 days or other vaccine within 14 days of vaccination;
* Receipt of blood transfusion or blood products 6 months prior to vaccination;
* Participation in another clinical study of an investigational product currently or within past 12 weeks or expected participation during this study;
* Receipt of another experimental HIV vaccine at any time;
* History of severe local or systemic reactogenicity to vaccination or history of severe allergic reactions;
* Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation in the previous 3 years;
* In the opinion of the investigator, unlikely to comply with protocol;
* ECG with clinically significant findings or features that would interfere with the assessment of myo/pericarditis including:
* conduction disturbance (atrioventricular or intraventricular condition, left or right bundle branch block, AV block of any degree, or QTc prolongation)
* repolarization (ST segment or T wave) abnormality
* significant atrial or ventricular arrhythmia
* frequent atrial or ventricular ectopy (e.g. frequent premature atrial contractions, 2 premature ventricular contractions in a row)
* ST elevation consistent with ischemia
* evidence of past or evolving myocardial infarction;

History of, or known active cardiac disease including:

* previous myocardial infarction (heart attack)
* angina pectoris
* congestive heart failure
* valvular heart disease including mitral valve prolapse
* cardiomyopathy
* pericarditis
* stroke or transient ischemic attack
* chest pain or shortness of breath with activity (such as walking up stairs)
* other heart conditions under the care of a doctor;

Have 3 or more of the following risk factors:

* high blood pressure diagnosed by a doctor
* high blood cholesterol diagnosed by a doctor
* diabetes or high blood sugar diagnosed by a doctor
* a first degree relative (for example, mother, father, brother, sister) who had a heart condition before the age of 50
* smoke cigarettes now.
* History of allergy to aminoglycosides (e.g. gentamycin)
* History of severe allergy to eggs or egg products e.g., "rash or breathing difficulties"

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of AMVA | 18 months

SECONDARY OUTCOMES:
Immunogenicity of ADMVA | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ho, MD, Principal Investigator — Aaron Diamond AIDS Research Center; Michael Keefer, MD, Principal Investigator — University of Rochester; Soe Than, MD, Study Director — International AIDS Vaccine Initiative
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Result] Vasan S, Schlesinger SJ, Chen Z, Hurley A, Lombardo A, Than S, Adesanya P, Bunce C, Boaz M, Boyle R, Sayeed E, Clark L, Dugin D, Boente-Carrera M, Schmidt C, Fang Q, LeiBa, Huang Y, Zaharatos GJ, Gardiner DF, Caskey M, Seamons L, Ho M, Dally L, Smith C, Cox J, Gill D, Gilmour J, Keefer MC, Fast P, Ho DD. Phase 1 safety and immunogenicity evaluation of ADMVA, a multigenic, modified vaccinia Ankara-HIV-1 B'/C candidate vaccine. PLoS One. 2010 Jan 25;5(1):e8816. doi: 10.1371/journal.pone.0008816. PMID 20111599
- [Derived] Elizaga ML, Vasan S, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One. 2013;8(1):e54407. doi: 10.1371/journal.pone.0054407. Epub 2013 Jan 17. PMID 23349878